CLINICAL TRIAL: NCT07132905
Title: Randomized Pilot Trial of Church-Based Problem-Solving Therapy for Adolescent Girls and Young Women With a History of Gender-Based Violence in Zambia
Brief Title: Mpata Yathu Trial for Young Women in Zambia
Acronym: MYT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-23-1685-AM-005; UCLA-CDU CFAR grant AI152501 (Other Grant/Funding Number: UCLA-CDU CFAR grant AI152501)
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: HIV; Common Mental Health Problems; PTSD - Post Traumatic Stress Disorder; Depression Disorder; Anxiety
Keywords: Gender-based violence; Problem-solving therapy; Adolescent girls and young women; Zambia; Lay counselors; Mental health; HIV treatment engagement; HIV prevention
MeSH Terms: conditions — Combat Disorders; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel assignment randomized controlled trial evaluating the effectiveness and implementation of Mpata Yathu, a church-based, lay counselor-delivered problem-solving therapy intervention for adolescent girls and young women (AGYW) in Zambia with a history of gender-based violence. Participants are randomized 1:1 to either an immediate intervention group (receiving six weekly PST sessions from baseline to 3 months) or a waitlist control group (receiving usual care from 0-3 months and the same intervention from 3-6 months). All participants are assessed at baseline, 3 months, and 6 months. The primary outcome is change in common mental disorder symptoms at 3 months. Implementation outcomes include feasibility, acceptability, and fidelity.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants and lay counselors delivering the intervention will not be blinded to study arm assignment. However, quantitative outcome assessors conducting follow-up assessments at 3 and 6 months will be blinded to participants' group assignment to reduce bias in data collection. These assessors will not participate in intervention delivery and will be trained to avoid accessing materials or communication that could reveal arm status. Unblinding will only occur in the event of an adverse event or safety concern requiring knowledge of the participant's group assignment for appropriate clinical referral or management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Mpata Yathu Intervention (Experimental): Participants randomized to this arm will receive the Mpata Yathu intervention immediately after enrollment. Mpata Yathu is a church-based, lay counselor-delivered adaptation of the Friendship Bench problem-solving therapy model. The intervention includes six weekly individual counseling sessions focused on structured problem-solving techniques and delivered in private spaces within local Catholic churches in Lusaka, Zambia. Counseling is provided by trained lay counselors who are pastors, teachers, peer navigators, and other trusted community members. Sessions are trauma-informed and survivor-centered, with integrated referrals for mental health, HIV, or GBV-related support services as needed. Follow-up assessments occur at 3 and 6 months.
  Interventions: Behavioral: Mpata Yathu ("Our Space")
- Waitlist Control - Delayed Mpata Yathu Intervention (Experimental): Participants in this arm will receive usual care during the first three months after enrollment and will then receive the Mpata Yathu intervention between Months 3 and 6. Mpata Yathu is a church-based, lay counselor-delivered problem-solving therapy adapted from the Friendship Bench model. It consists of six weekly individual counseling sessions, delivered in church settings by trained lay counselors using a trauma-informed, survivor-centered approach. Sessions include structured problem-solving and optional referrals for HIV, GBV, or mental health services. Follow-up assessments are conducted at 3 months (pre-intervention) and again at 6 months (post-intervention).
  Interventions: Behavioral: Mpata Yathu ("Our Space")

INTERVENTIONS:
Behavioral: Mpata Yathu ("Our Space") — Mpata Yathu is a church-based, lay counselor-delivered psychological intervention adapted from the Friendship Bench problem-solving therapy (PST) model. Designed for adolescent girls and young women in Zambia with a history of gender-based violence and elevated mental health symptoms, the intervention includes six weekly individual PST sessions delivered in private spaces within Catholic churches. Lay counselors are trained in trauma-informed, survivor-centered care and offer optional referrals to mental health, HIV, or GBV-related services. Mpata Yathu maintains the core structure of Friendship Bench but was adapted through community-partnered participatory research to meet the sociocultural needs of Zambian youth.
  Other Names: Church-Based Problem-Solving Therapy; Lay counselor-delivered Problem-Solving Therapy

SUMMARY:
This study aims to improve mental health and HIV-related outcomes among adolescent girls and young women (AGYW) in Zambia who have experienced gender-based violence (GBV). GBV includes physical, sexual, or emotional violence from partners or others and is known to increase the risk of depression, anxiety, post-traumatic stress, and HIV infection. In Zambia, access to mental health services is limited, especially for young women in low-resource communities. This study tests a counseling program called Mpata Yathu, which means "Our Space" in Chinyanja, designed to provide psychological support and improve well-being for young women who have faced violence and may be living with or at risk for HIV.

Mpata Yathu is a culturally adapted version of the Friendship Bench, a lay counselor-delivered mental health intervention originally developed in Zimbabwe. In this adapted version, trained community lay counselors will deliver six individual problem-solving therapy (PST) sessions over a three-month period. Sessions will be delivered in private spaces within local Catholic churches in the Matero and Chawama areas of Lusaka, Zambia. Counseling sessions will also include referral options for participants who may need further support related to HIV care, GBV, or mental health concerns.

The study is a two-arm randomized controlled trial. Participants will be randomly assigned to either:

1. Immediate Intervention Group - Receives the Mpata Yathu intervention between baseline and 3-month follow-up
2. Waitlist Control Group - Receives usual care for the first 3 months and then receives the Mpata Yathu intervention between 3- and 6-month follow-up

A total of 180 young women (90 per group) will participate in the trial. To be eligible, participants must be between the ages of 15 and 24, reside in the Matero or Chawama area, report lifetime GBV exposure, and show moderate depressive symptoms or symptoms of common mental disorders (CMDs). They must also be living with HIV or report behaviors that place them at risk for HIV.

The primary outcome is symptoms of CMDs, assessed using the Shona Symptom Questionnaire (SSQ-14). Secondary outcomes include depression, anxiety, and PTSD symptoms, as well as HIV-related outcomes such as clinic attendance, antiretroviral therapy (ART) adherence, and prevention behaviors such as condom use or PrEP readiness. The study will also measure feasibility, acceptability, and fidelity of the intervention.

Data will be collected through surveys at baseline, 3 months, and 6 months. The research team will also monitor how the intervention is implemented, how participants respond to counseling, and whether counselors follow the therapy protocol. Participants will receive a small stipend for their time and transport at each counseling session and follow-up visit.

This study is designed to test whether a trauma-informed, church-based mental health intervention can improve psychological well-being and HIV engagement among young women who are often underserved in traditional healthcare systems. If successful, this model could be expanded to other churches or schools in Zambia and similar settings. The results will inform future large-scale evaluations and could help shape new strategies for addressing GBV, mental health, and HIV among youth in sub-Saharan Africa.

DETAILED DESCRIPTION:
Background

Young women, aged 15 to 24 years, in Zambia are vulnerable to gender-based violence (GBV)1 such as intimate partner violence (IPV), forced sex, other forms of sexual assault, and stalking. GBV increases risks for HIV acquisition by 50% in high HIV-burden countries like Zambia. The HIV prevalence among Zambian young women is three times higher than their male counterparts and positive HIV status among these women is significantly associated with experiencing IPV. GBV-exposed women are also at elevated risk for mental health disorders (depression, anxiety, PTSD, substance abuse). In a cohort study of 1,915 young women in Zambia, women who experienced sexual violence perpetrated by non-partners had increased odds of depression and anxiety. GBV and mental health disorders also undermine HIV prevention and treatment including antiretroviral therapy adherence, clinic attendance, and pre-exposure prophylaxis (PrEP) use. Young Zambians who have experienced physical violence, psychological abuse, or forced sex have higher odds of HIV viral load suppression failure. Although the integration of mental health treatments within HIV interventions can lead to improvements in HIV and mental health outcomes, there is insufficient evidence of this impact among young women with a history of GBV in low-resource settings like Zambia. Therefore, we propose to pilot test the integration of a locally adapted, lay-delivered evidence-based problem solving therapy intervention, known as Mpata Yathu, to improve mental health and HIV prevention and treatment outcomes among young women with a history of GBV in Zambia. This protocol outlines the evaluation of Mpata Yathu, which aims to:

1. Assess the effect of the intervention on common mental health disorder (CMD) symptoms, the primary outcome for which the study is statistically powered.
2. Evaluate the implementation outcomes of the Mpata Yathu intervention, specifically its feasibility, acceptability, and fidelity, as delivered by lay counselors to AGYW with a history of GBV experiences.
3. Explore potential effects of the Mpata Yathu intervention on additional mental health outcomes such as depression, anxiety, and PTSD; HIV prevention and treatment engagement outcomes based on participant HIV status; and gender-based violence (GBV)-related attitudes and experiences, as well as psychosocial variables including adverse childhood experiences and coping self-efficacy.
4. Whether changes in mental health symptoms mediate or moderate the intervention's effects on HIV-related outcomes.

Methods

Study Design We will conduct a two-arm randomized controlled trial (RCT) to evaluate the effectiveness and implementation of the adapted Friendship Bench intervention, Mpata Yathu, on HIV prevention and treatment, and depression outcomes among young women, living with or at risk for HIV, with a lifetime history of GBV and depression symptoms in Zambia. This study will have two arms: an intervention group and a waitlist control group. The intervention is designed to be delivered in six sessions, with one session per week. However, participants will be given up to three months to complete all sessions to accommodate common barriers such as caregiving responsibilities, stigma, mobility, and illness. Counseling sessions will be scheduled to accommodate participant availability, and lay counselors will track session completion. After screening and enrollment, eligible participants will be randomized in a 1:1 ratio to either group.

Intervention Group: Participants will receive up to six individual counseling sessions between baseline and 3-month follow-up (0-3 months).

Waitlist Control Group: Participants will receive usual care from 0-3 months, followed by the intervention (up to six counseling sessions) between 3 and 6 months

Due to the nature of the intervention, participants and lay counselors will not be blinded to study arm assignment. However, quantitative outcome assessors conducting follow-up assessments will be blinded to participants' group assignment to reduce potential bias in data collection. Unblinding will only occur in cases of adverse events or safety concerns where knowledge of intervention status is necessary for appropriate clinical management or referral.

Study Setting Our study will be conducted in two Roman Catholic churches in Lusaka, one located in the Matero catchment area and one located in Chawama. Our community partners, who are Native Zambians, recommended implementation of Friendship Bench within churches in the Matero and Chawama catchment areas of Lusaka since women are disproportionately affected by both poverty and GBV in these areas, aligning with literature linking economic vulnerability to sexual coercion. Roman Catholic churches were recommended by native Zambians as appropriate sites for implementation since they serve a wide population and offer the classroom space and organizational structure needed to host counseling sessions.

Screening and Enrollment We anticipate screening 300 young women over four months to enroll 90 eligible participants. We are planning for a conservative dropout rate of 30%. This estimate draws from comparable implementation research in sub-Saharan Africa, including a trial in rural Ethiopia, which used a similar assumption to test feasibility of participant retention and study procedures. This estimate allows us to account for structural barriers (e.g., mobility, stigma, early pregnancy, GBV recurrence, financial hardship, caregiving responsibilities) that commonly affect longitudinal follow-up among AGYW who have experienced GBV. Collecting actual retention data during the RCT will allow us to empirically estimate the true dropout rate and its variability, which will inform the design and sample size calculations of a future fully powered randomized controlled trial, and for refining strategies to improve participant retention.

Participants will be considered lost to follow-up for a specific assessment (at 3 or 6 months after the baseline assessment) if they cannot be reached despite at least three documented re-contact attempts using various methods (e.g., phone calls, church-based outreach, or home visits, based on participant consent and preference) during the assessment window, defined as ±1 month from the target follow-up date. Re-contact efforts will begin approximately two weeks prior to each window and continue throughout. No outreach will occur after the close of each window. Participants who miss the 3-month follow-up assessment may still be contacted and retained for the 6-month follow-up. Participants who voluntarily withdraw from the study will not be considered lost to follow-up.

Randomization We will use permuted block randomization, stratified by HIV status, to ensure balance across study arms. The randomization sequence will be computer-generated using REDCap's randomization module. REDCap will conceal allocation until after baseline data entry is complete, ensuring that research staff cannot foresee or manipulate assignments. The study biostatistician will generate the allocation sequence and upload it into REDCap. The research assistants will enroll participants, and REDCap will automatically assign the participant to their group after enrollment and baseline data completion. Participants will be randomized 1:1 to the intervention group (offering intervention sessions from 0-3 months) or the waitlist control group (offering intervention sessions from 3-6 months), with up to six sessions delivered over three months among both arms.

Inclusion Criteria

To be eligible for enrollment in the RCT, participants must meet the following criteria:

1. aged 15 to 24 years;
2. Speak Nyanja, Bemba, and/or English fluently;
3. Reside in the Matero or Chawama constituency area during the time of recruitment;
4. Report lifetime exposure to GBV, as assessed by the WHO Multi-country Study on Women's Health and Domestic Violence Against Women instrument.
5. Exhibit moderate depressive symptoms indicated by a score of 10-14 on the 9-item Patient Health Questionnaire (PHQ-9), or common mental disorder (CMD) symptoms (e.g., depression, anxiety) as indicated by a score of 9 or higher on the 14-item Shona Symptom Questionnaire (SSQ-14); and
6. Be living with HIV or demonstrate HIV risk behaviors, as defined by validated items from the World AIDS Foundation survey, including unprotected sex, multiple sexual partners, coerced sex, or transactional sex.

Exclusion Criteria

Women will be excluded if they:

1. Require emergency treatment for any crisis (mental, physical, emotional) at the time of screening
2. Report severe symptoms of depression (score > 14 on PHQ-9) or no to mild depression symptoms (PHQ-9 score <10), and/or severe anxiety symptoms using the Generalized Anxiety Disorder 7-item scale or GAD-7 (score >14 on GAD-7)
3. Have intellectual or cognitive disabilities that limit their ability to complete the screening tools, interact with a lay counselor and/or provide informed consent; and/or
4. Are considered in immediate danger (e.g., reoccurring physical violence) during time of the study.
5. Are currently receiving formal mental health counseling or psychotherapy (to avoid duplication of care and potential confounding effects).

Study Procedures for RCT Participants Recruitment, screening, and consenting will take place at both intervention and non-intervention sites across Lusaka, including churches, government health facilities, schools, and community-based organizations; the intervention will be delivered at two Catholic churches-one in Matero and the other in Chawama. These locations were identified in consultation with native Zambians who are familiar with these church settings to ensure accessibility and safety for potential participants. Private rooms within the selected locations will be used to ensure confidentiality during screening and consenting. In some cases where private rooms are unavailable, screening and consenting will take place outdoors in quiet, secluded areas to maintain privacy.

Participants will be informed whether they are eligible for the study immediately after completing the screening. Eligible individuals will be considered enrolled in the study immediately after consenting. If unavailable to screen, consent, and/or enroll during the time of recruitment, potential participants will be asked to schedule a time to complete the screening, enrolling, and/or consenting in person.

Consenting will be conducted by the local study team, including pastors, students, teachers, and youth peer navigators, who have completed training in research ethics and informed consent procedures. While some lay counselors delivering the intervention may also assist with consenting, they will not administer baseline or follow-up questionnaires to avoid potential bias in participant responses. All study personnel, including the lay counselors, will be certified in human subjects protection prior to study launch and follow safety protocols for women who may still be experiencing GBV and/or have specific mental health needs outside of the scope of our study (e.g., severe depression, suicidal ideation or attempt, psychosis).

Study Outcomes All outcomes will be assessed at both 3-month and 6-month follow-up timepoints. The 3-month follow-up will serve as the primary endpoint for between-group comparisons (intervention vs. waitlist control). At the 6-month follow-up, only within-group changes will be assessed, as both groups will have received the intervention by this time. The waitlist control group will begin intervention delivery after completing the 3-month assessment, with no contamination expected due to the ±1 month window applied to the time in which follow-up assessments must be completed. All instruments will be translated into from English to Nyanja and Bemba using a forward-backward translation process to ensure linguistic and cultural equivalence.

Mental Health Outcomes The primary outcome is symptoms of common mental disorders (CMDs), assessed using the Shona Symptom Questionnaire (SSQ-14). The SSQ-14 consists of 14 yes/no items assessing psychological distress, with a score ≥9 indicating probable CMD. This outcome will be measured at 3 months and analyzed as a continuous variable, consistent with the original Friendship Bench study, which used SSQ-14 scores as a continuous measure to assess symptom reduction overtime. The SSQ-14 was selected as the primary outcome measure because it is a culturally adapted and validated screening tool developed specifically for Zimbabwean and similar Southern African primary care populations. It captures symptoms of CMDs across emotional, somatic, and functional domains, and demonstrated strong psychometric properties in the original Friendship Bench trial.

The secondary outcome is depressive symptoms, measured using the Patient Health Questionnaire-9 (PHQ-9). PHQ-9 scores will also be analyzed using both binary and continuous analysis, consistent with the original Friendship Bench trial.26 Although eligibility for this study includes a PHQ-9 score between 10-14, PHQ-9 will also be analyzed as a binary variable using a cutoff of ≥11 to estimate the prevalence of probable depression, as done in the original trial. The PHQ-9 was selected as the secondary outcome due to its global recognition and its use in clinical settings in Zambia. Using the PHQ-9 enables broader comparability with global mental health studies and potential clinical integration. Exploratory mental health outcomes include anxiety and PTSD symptoms, assessed with the Generalized Anxiety Disorder (GAD-7) scale and Child PTSD Symptom Scale (CPSS), respectively. CPPS was validated among children and adolescents in Zambia with good internal reliability (α>.80).

HIV Outcomes All HIV-related outcomes (treatment and prevention) are exploratory but will be measured at baseline and at 3- and 6-month follow-up. We will assess HIV prevention engagement and risk behaviors among participants in our study that are not living with HIV, using a self-reported survey on HIV risk behaviors using measures from the World AIDS Foundation (WAF) Survey. We will also administer the HIV Prevention Readiness Measure (HPRM)65 at both baseline and follow-up. The HPRM is a validated instrument originally developed for the HPTN 082 study to assess readiness for and sustained use of HIV prevention strategies such as PrEP among AGYW in sub-Saharan Africa. It includes subscales on self-efficacy, disclosure, and social support, which are strong indicators of behavioral and psychosocial engagement in HIV prevention.

HIV treatment engagement will be assessed among participants living with HIV through both self-reported and clinical measures. We will distinguish between women who are already diagnosed with HIV and those who may be newly diagnosed during the study period. For women already diagnosed with HIV, we will assess self-reported clinic attendance over the past 6 months, recognizing that visit frequency may vary by treatment regimen and differentiated service delivery model (e.g., 1-, 3-, or 6-month refill cycles). Where available, participants will be asked to voluntarily share their health passport or personal medical record to assess additional treatment engagement indicators such as their most recent HIV viral load, ART regimen, pharmacy refills or missed doses (if noted), and clinic attendance.For women newly diagnosed during the study, we will use the following engagement indicators to assess initial linkage to care: the date and location of their most recent HIV test; whether and where they linked to a clinic or facility for confirmatory testing and care; whether they were referred to care by a member of the study team; and whether ART was initiated, including how soon after diagnosis it began. Lastly, HIV treatment self-efficacy among seropositive participants will be assessed using the HIV Self-Efficacy Questionnaire (HIV-SE), which reflects participants' confidence in managing their HIV care and may be correlated with treatment engagement.

GBV Experiences, Attitudes, and Perceptions GBV-related experiences, attitudes and perceptions will be measured as exploratory outcomes. Experiences of GBV will be assessed using the WHO Multi-country Study on Women's Health and Domestic Violence Against Women Instrument2 (Sections 7-10: physical, sexual, and emotional violence by partners and non-partners), while attitudes and risk perceptions will be evaluated using Section 6 of the same instrument. GBV perceptions will also be measured using Perrin et al.'s Social Norms and Beliefs about Gender-Based Violence Scale.67 These measures were selected for their strong psychometric properties and relevance to sub-Saharan African contexts. Including both experience- and perception-based measures will allow us to assess participants' attitudes and beliefs, which may serve as important indicators of GBV risk.

Implementation Outcomes We will quantitatively assess feasibility outcomes, acceptability, and fidelity. Acceptability will be measured by evaluating retention rate (i.e., number of participants and lay counselors who drop out of the intervention) and safety (i.e., number of adverse events reported to the Institutional Review Board). To assess the acceptability of the intervention from the perspective of participants, we will use the Acceptability of Intervention Measure. AIM is a 4-item scale that captures participants' overall perceptions of the intervention's acceptability, using a 5-point Likert response format. These items assess whether participants found the intervention appealing, satisfactory, and appropriate. Acceptability will also be measured through semi-structured interviews with participants and lay counselors as described below. This mixed-method approach (close- and open-ended items) will provide both quantitative and qualitative data on acceptability and identify areas for improvement in future implementation.

Lay counselor adherence to the protocol will be monitored using a fidelity checklist and weekly supervision sessions. Fidelity will capture lay counselors' adherence to core problem-solving therapy techniques. Fidelity will be assessed through audio recordings of counseling sessions, contingent upon participant consent, as individuals may choose to opt out of being recorded. During the initial phase of implementation (within the first two weeks), all the sessions will be reviewed in a timely manner to provide formative feedback and support counselor development. A random sample of approximately 20% of recorded sessions will be evaluated thereafter.

Lastly, we will qualitatively assess barriers and facilitators of Friendship Bench implementation via semi-structured interviews on intervention experiences among study participants and lay counselors using relevant domains and constructs from the Consolidated Framework for Implementation Research (CFIR), and the modified CFIR for LMICs. We are hoping that capturing barriers and facilitators would also allow us to qualitatively assess satisfaction and burden (i.e., risks and benefits associated with participation among counselors and clients). We will qualitatively assess the feasibility and acceptability of the intervention through semi-structured interviews with both participants and lay counselors. All lay counselors who delivered the intervention (up to 12 total) will be invited to voluntarily participate in an interview. Additionally, we will conduct up to 15 interviews with participants from each study arm (intervention and delayed control group) to gather diverse perspectives on the intervention experience. To accommodate participants who are not fluent or comfortable communicating in English, interviews will be conducted in local languages (e.g., Nyanja or Bemba) by trained bilingual interviewers. All audio recordings will be transcribed and then translated into English (if applicable) for analysis. To ensure accuracy and cultural validity, a subset of transcripts will undergo back-translation and review by the research team.

We will also qualitatively evaluate content coverage of sessions which will include documentation of whether counselors explore topics such as interpersonal challenges (e.g., family or peer relationships), past (not current) experiences of violence, suicidal ideation or distress, and HIV treatment or prevention challenges. These areas are consistent with known stressors among the target population and align with the intervention's goals of improving coping and mental health outcomes. Content coverage will be assessed as a process measure (i.e., what topics came up in sessions), and as an implementation determinant (i.e., why some topics were avoided or emphasized), especially based on lay counselor interviews or debriefs.

Participant responsiveness will be qualitatively assessed through multiple sources. First, we will conduct semi-structured interviews with both lay counselors and participants to explore how participants experienced the Friendship Bench sessions, which may give us insight on their level of engagement, perceived relevance of the content, and emotional or behavioral reactions. Second, we will analyze post-session summary notes completed by lay counselors after each session, which include reflections on how engaged the participant appeared, whether they participated in problem-solving activities, and how they responded to the session content. Additionally, study team debrief notes-documenting informal observations and key discussion points during supervision meetings-will be reviewed to triangulate findings and assess patterns of responsiveness across participants. This multi-source, qualitative approach will provide a rich understanding of participant responsiveness and help inform adaptations to enhance engagement in future implementation.

Psychosocial Outcomes All psychosocial measures are exploratory. We will include the Adverse Childhood Experiences International Questionnaire (ACE-IQ) and the Coping Self-Efficacy (CSE) scale as exploratory psychosocial measures. The ACE-IQ assesses exposure to early life adversity, providing context for participants' mental health needs and potential barriers to care. The CSE scale measures perceived ability to cope with stress through problem-solving, emotional regulation, and social support. Lastly, we will be measuring social support using the 3-item Oslo social support scale (OSSS-3), which measure the number of close confidants, perceived concern from others, and ease of obtaining practical help. Together, these tools will help us explore how early adversity and coping capacity may influence engagement with the intervention and inform future trauma- and resilience-informed adaptations.

Power Analysis This RCT is powered only to detect intervention effects on symptoms of CMDs, as measured by the SSQ-14, which is the primary outcome. All other quantitative outcomes-including other mental health measures, HIV engagement indicators, and psychosocial variables-will be treated as exploratory and used to inform effect size estimates and future trial design. With the proposed sample size of 180 participants (90 per arm) and using a two-sided alpha level of 0.05, the study will have 80% power to detect a medium effect size of Cohen's d = 0.5 in SSQ-14 scores, which will be analyzed as a continuous outcome. This is a conservative estimate, selected to reflect a clinically meaningful but smaller effect than that observed in the original Friendship Bench trial, which reported a large effect (d ≈ 0.75-0.8) over a 6-month period. Since our study primarily measures outcomes at 3 months, a smaller effect size is assumed to avoid overestimating power. Between-group comparisons will be conducted at the 3-month follow-up, prior to the waitlist control group receiving the intervention. At 6 months, only within-group analyses will be conducted to assess sustained changes in the intervention group and pre-post change in the waitlist control group. No between-group comparisons will be performed at 6 months.

Quantitative Data Analysis We will use descriptive statistics to summarize participant characteristics at baseline, feasibility and acceptability metrics, and other implementation outcomes. To assess baseline differences between participants who complete the intervention and those who drop out, we will conduct bivariate comparisons using independent samples t-tests or Wilcoxon rank-sum tests for continuous variables, and chi-square or Fisher's exact tests for categorical variables.

Primary Outcome Analysis (Powered): To assess the effect of the adapted intervention on symptoms of CMDs (SSQ-14), we will use mixed-effects linear regression models. This is the only outcome for which the study is statistically powered, based on detecting a standardized mean difference of Cohen's d = 0.5 at the 3-month follow-up.

Exploratory Analyses: All other outcomes will be analyzed using mixed-effects linear, logistic, or ordinal regression models, depending on the outcome type. These outcomes include mental health outcomes, HIV prevention outcomes, HIV treatment outcomes, and HIV treatment self-efficacy.

Moderation and Mediation Analyses (Exploratory): Post-hoc exploratory analyses will assess whether changes in mental health outcomes mediate or moderate the intervention's effects on HIV-related outcomes. Mental health change scores will be calculated separately for each follow-up period (i.e., 3 months and 6 months post-intervention) by subtracting baseline values from the respective follow-up values. This will allow us to assess both short-term and sustained mental health changes and explore their relationship with HIV-related outcomes over time.

Adjustment Variables and Stratified Analyses: HIV status (positive vs. negative/unknown) will be included as a covariate in pooled models to adjust for baseline differences. Stratified analyses by HIV status will be considered if each group has a sufficient sample size to support reliable subgroup modeling (e.g., ≥40 participants per group). Given the small overall sample size (N = 90, accounting for 30% attrition), such stratified analyses may be underpowered and are therefore considered exploratory and hypothesis-generating only. All models will follow an intention-to-treat framework, and statistical significance will be assessed at a two-sided α = 0.05, with 95% confidence intervals reported.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment in the RCT, participants must meet the following criteria:

1. aged 15 to 24 years;
2. Speak Nyanja, Bemba, and/or English fluently;
3. Reside in the Matero or Chawama constituency area during the time of recruitment;
4. Report lifetime exposure to GBV, as assessed by the following sections of the WHO Multi-country Study on Women's Health and Domestic Violence Against Women instrument:

   * Section 7 (Physical Violence by Intimate Partner): Reports of being slapped, pushed, hit with a fist, kicked, dragged, choked, or threatened/attacked with a weapon by a husband or partner.
   * Section 8 (Sexual Violence by Intimate Partner): Reports of being physically forced to have sex, having sex out of fear, or being forced to engage in degrading sexual acts by a husband or partner.
   * Section 9 (Emotional Abuse by Intimate Partner): Reports of being insulted, belittled, intimidated, or threatened by a partner.
   * Section 10 (Physical Violence by Non-Partner): Lifetime experiences of being beaten or physically mistreated by someone other than a partner since age 15.
   * Section 11 (Sexual Violence by Non-Partner): Forced sex or sexual acts since age 15 by a non-partner, and childhood sexual abuse before age 15.
5. Exhibit moderate depressive symptoms indicated by a score of 10-14 on the 9-item Patient Health Questionnaire (PHQ-9), or common mental disorder (CMD) symptoms (e.g., depression, anxiety) as indicated by a score of 9 or higher on the 14-item Shona Symptom Questionnaire (SSQ-14); and
6. Be living with HIV or demonstrate HIV risk behaviors, as defined by validated items from the World AIDS Foundation survey,25 including unprotected sex, multiple sexual partners, coerced sex, or transactional sex.

Exclusion Criteria:

Women will be excluded if they:

1. Require emergency treatment for any crisis (mental, physical, emotional) at the time of screening
2. Report severe symptoms of depression (score > 14 on PHQ-9) or no to mild depression symptoms (PHQ-9 score <10), and/or severe anxiety symptoms using the Generalized Anxiety Disorder 7-item scale or GAD-7 (score >14 on GAD-7)
3. Have intellectual or cognitive disabilities that limit their ability to complete the screening tools, interact with a lay counselor and/or provide informed consent; and/or
4. Are considered in immediate danger (e.g., reoccurring physical violence) during time of the study.
5. Are currently receiving formal mental health counseling or psychotherapy (to avoid duplication of care and potential confounding effects).

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This study is limited to individuals who self-identify as female. Eligible participants must be adolescent girls and young women aged 15 to 24 who identify as female, regardless of their assigned sex at birth. Individuals of other gender identities are not eligible for this study.
Enrollment: 180 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of common mental disorders (CMDs) as measured by the Shona Symptom Questionnaire (SSQ-14) | Baseline and 3-month follow-up
  The primary outcome is change in symptoms of common mental disorders (CMDs), measured using the Shona Symptom Questionnaire (SSQ-14), a 14-item screening tool used in Friendship Bench studies. Each item is scored as 0 or 1, with a total score range of 0-14. Higher scores reflect greater symptom severity. The primary analysis will compare mean SSQ-14 scores between the intervention and waitlist control arms at the 3-month follow-up, prior to the waitlist group receiving the intervention. SSQ-14 will also be measured at 6 months to assess within-group changes, but this is not part of the primary between-group analysis.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3-month, and 6-month follow-up
  Depressive symptoms will be assessed using the 9-item Patient Health Questionnaire (PHQ-9), a widely used and validated screening tool for depression. Each item is scored from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27. Higher scores indicate more severe depressive symptoms. Mean PHQ-9 scores will be compared between arms at 3-month follow-up, with additional within-group change explored at 6-month follow-up.
Change in anxiety symptoms as measured by the Generalized Anxiety Disorder-7 (GAD-7) scale | Baseline, 3-month, and 6-month follow-up
  Anxiety symptoms will be measured using the 7-item GAD-7 scale. Each item is scored on a 0-3 scale, with a total possible score of 21. Higher scores reflect more severe anxiety symptoms. Mean scores will be compared across arms at 3-month follow-up and assessed for within-group change at 6 months.
Change in PTSD symptoms as measured by the Child PTSD Symptom Scale (CPSS) | Baseline, 3-month, and 6-month follow-up
  PTSD symptoms will be measured using the Child PTSD Symptom Scale (CPSS), a 24-item self-report instrument designed to assess post-traumatic stress symptoms and related functional impairments in adolescents. The scale includes 17 items corresponding to DSM-IV PTSD symptom criteria and 7 items assessing functional impairment in areas such as school, family, and social life. Each symptom item is scored from 0 (not at all) to 3 (5 or more times a week), with a total symptom severity score ranging from 0 to 51. Scores will be compared between groups at 3-month follow-up, and within groups at 6-month follow-up.

OTHER OUTCOMES:
HIV treatment engagement among participants living with HIV | Baseline, 3-month, and 6-month follow-up
  Among participants living with HIV, treatment engagement will be assessed using self-reported clinic attendance and, where available, clinical data such as viral load, ART regimen, and pharmacy refills. Data will be collected at each follow-up to explore whether participation in Mpata Yathu is associated with improved treatment engagement. This outcome is exploratory and not powered for hypothesis testing.
HIV prevention readiness and behaviors among participants at risk for HIV | Baseline, 3-month, and 6-month follow-up
  Among HIV-negative participants, HIV prevention readiness and behaviors will be assessed using survey questions on condom use, HIV testing, prevention self-efficacy, and PrEP awareness/readiness. Changes over time will be examined to explore potential effects of the Mpata Yathu intervention. This is an exploratory outcome.
Attitudes toward gender-based violence (GBV) and recent GBV experiences | Baseline, 3-month, and 6-month follow-up
  Participants will complete validated measures assessing attitudes toward GBV, social norms, and recent experiences of emotional, physical, or sexual violence. These data will help explore whether Mpata Yathu influences GBV-related beliefs and exposures. This outcome is exploratory.
Change in coping self-efficacy as measured by the Coping Self-Efficacy Scale (CSE) | Baseline, 3-month, and 6-month follow-up
  The CSE Scale assesses confidence in managing stress, emotions, and problem-solving. Items are scored 0-10, with higher scores indicating stronger coping ability. This exploratory outcome will be used to assess potential psychosocial changes resulting from the intervention.
Perceived social support as measured by the Oslo Social Support Scale (OSS-3) | Baseline, 3-month, and 6-month follow-up
  The OSS-3 is a 3-item scale measuring the availability and perceived adequacy of social support. Scores range from 3 to 14. This outcome will be used to explore whether the Mpata Yathu intervention affects social support among participants.

CONTACTS AND LOCATIONS:
Overall Officials: Charisse V Ahmed, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Not applicable (multi-site study), Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual-level quantitative data collected through participant surveys, including responses to validated mental health, HIV, GBV, and psychosocial measures, will be shared. No identifying information such as names, contact details, or GPS coordinates will be included. Audio recordings and qualitative interview transcripts will not be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified IPD and supporting materials will be made available beginning 12 months after primary publication. Data will remain accessible indefinitely, as long as the Principal Investigator and study team are able to maintain secure and ethical data sharing processes. Access will be granted upon review of data access requests and completion of required approvals and agreements.
Access Criteria: Data will be available to researchers with a methodologically sound proposal, subject to approval by the Principal Investigator and study team. Requestors must submit a data access application outlining research aims and methods. Access will be granted through a secure data-sharing platform or encrypted transfer, contingent on ethical approvals and signed data use agreements. Data will be de-identified to protect participant confidentiality.

REFERENCES:
- [Background] White SJ, Sin J, Sweeney A, Salisbury T, Wahlich C, Montesinos Guevara CM, Gillard S, Brett E, Allwright L, Iqbal N, Khan A, Perot C, Marks J, Mantovani N. Global Prevalence and Mental Health Outcomes of Intimate Partner Violence Among Women: A Systematic Review and Meta-Analysis. Trauma Violence Abuse. 2024 Jan;25(1):494-511. doi: 10.1177/15248380231155529. Epub 2023 Feb 24. PMID 36825800
- [Background] Stein C, Flor LS, Gil GF, Khalil M, Herbert M, Aravkin AY, Arrieta A, Baeza de Robba MJ, Bustreo F, Cagney J, Calderon-Anyosa RJC, Carr S, Chandan JK, Chandan JS, Coll CVN, de Andrade FMD, de Andrade GN, Debure AN, DeGraw E, Hammond B, Hay SI, Knaul FM, Lim RQH, McLaughlin SA, Metheny N, Minhas S, Mohr JK, Mullany EC, Murray CJL, O'Connell EM, Patwardhan V, Reinach S, Scott D, Spencer CN, Sorensen RJD, Stockl H, Twalibu A, Valikhanova A, Vasconcelos N, Zheng P, Gakidou E. The health effects associated with physical, sexual and psychological gender-based violence against men and women: a Burden of Proof study. Nat Hum Behav. 2025 Jun;9(6):1201-1216. doi: 10.1038/s41562-025-02144-2. Epub 2025 Apr 10. PMID 40210704
- [Background] Kuchukhidze S, Panagiotoglou D, Boily MC, Diabate S, Eaton JW, Mbofana F, Sardinha L, Schrubbe L, Stockl H, Wanyenze RK, Maheu-Giroux M. The effects of intimate partner violence on women's risk of HIV acquisition and engagement in the HIV treatment and care cascade: a pooled analysis of nationally representative surveys in sub-Saharan Africa. Lancet HIV. 2023 Feb;10(2):e107-e117. doi: 10.1016/S2352-3018(22)00305-8. Epub 2022 Dec 1. PMID 36463914
- [Background] Ahmed C, Thornicroft M, Ntebeka BM, Chileshe, K, et al. Church-Based Problem-Solving Therapy for Adolescent Girls and Young Women with a History of Gender-Based Violence in Zambia: Study Protocol for a Hybrid Type 1 Randomized Controlled Trial. 2025 Jul 8. PREPRINT (Version 1) available at Research Square. https://doi.org/10.21203/rs.3.rs-7039714/v1
- [Background] Means AR, Kemp CG, Gwayi-Chore MC, Gimbel S, Soi C, Sherr K, Wagenaar BH, Wasserheit JN, Weiner BJ. Evaluating and optimizing the consolidated framework for implementation research (CFIR) for use in low- and middle-income countries: a systematic review. Implement Sci. 2020 Mar 12;15(1):17. doi: 10.1186/s13012-020-0977-0. PMID 32164692
- [Background] Dworkin ER, Weaver TL. The impact of sociocultural contexts on mental health following sexual violence: A conceptual model. Psychol Violence. 2021 Sep;11(5):476-487. doi: 10.1037/vio0000350. PMID 34631201
- [Background] Li Y, Marshall CM, Rees HC, Nunez A, Ezeanolue EE, Ehiri JE. Intimate partner violence and HIV infection among women: a systematic review and meta-analysis. J Int AIDS Soc. 2014 Feb 13;17(1):18845. doi: 10.7448/IAS.17.1.18845. eCollection 2014. PMID 24560342
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Chibanda D, Mesu P, Kajawu L, Cowan F, Araya R, Abas MA. Problem-solving therapy for depression and common mental disorders in Zimbabwe: piloting a task-shifting primary mental health care intervention in a population with a high prevalence of people living with HIV. BMC Public Health. 2011 Oct 26;11:828. doi: 10.1186/1471-2458-11-828. PMID 22029430
- [Background] Maddoux J, Symes L, McFarlane J, Koci A, Gilroy H, Fredland N. Problem-solving and mental health outcomes of women and children in the wake of intimate partner violence. J Environ Public Health. 2014;2014:708198. doi: 10.1155/2014/708198. Epub 2014 Nov 11. PMID 25435885
- [Background] Devries KM, Mak JY, Bacchus LJ, Child JC, Falder G, Petzold M, Astbury J, Watts CH. Intimate partner violence and incident depressive symptoms and suicide attempts: a systematic review of longitudinal studies. PLoS Med. 2013;10(5):e1001439. doi: 10.1371/journal.pmed.1001439. Epub 2013 May 7. PMID 23671407
- [Background] Conroy AA, Jain JP, Sheira L, Frongillo EA, Neilands TB, Cohen MH, Wilson TE, Chandran A, Adimora AA, Kassaye S, Sheth AN, Fischl MA, Adedimeji A, Turan JM, Tien PC, Weiser SD. Mental Health Mediates the Association Between Gender-Based Violence and HIV Treatment Engagement in US Women. J Acquir Immune Defic Syndr. 2022 Feb 1;89(2):151-158. doi: 10.1097/QAI.0000000000002848. PMID 34723926
- [Background] Leddy AM, Weiss E, Yam E, Pulerwitz J. Gender-based violence and engagement in biomedical HIV prevention, care and treatment: a scoping review. BMC Public Health. 2019 Jul 8;19(1):897. doi: 10.1186/s12889-019-7192-4. PMID 31286914
- [Background] Cabral A, M Baeten J, Ngure K, Velloza J, Odoyo J, E Haberer J, Celum C, Muwonge T, Asiimwe S, Heffron R; Partners Demonstration Project Team. Intimate Partner Violence and Self-Reported Pre-exposure Prophylaxis Interruptions Among HIV-Negative Partners in HIV Serodiscordant Couples in Kenya and Uganda. J Acquir Immune Defic Syndr. 2018 Feb 1;77(2):154-159. doi: 10.1097/QAI.0000000000001574. PMID 29076883
- [Background] Cluver L, Meinck F, Toska E, Orkin FM, Hodes R, Sherr L. Multitype violence exposures and adolescent antiretroviral nonadherence in South Africa. AIDS. 2018 May 15;32(8):975-983. doi: 10.1097/QAD.0000000000001795. PMID 29547438
- [Background] Merrill KG, Campbell JC, Decker MR, McGready J, Burke VM, Mwansa JK, Miti S, Frimpong C, Kennedy CE, Denison JA. Past-Year Violence Victimization is Associated with Viral Load Failure Among HIV-Positive Adolescents and Young Adults. AIDS Behav. 2021 May;25(5):1373-1383. doi: 10.1007/s10461-020-02958-3. PMID 32761474
- [Background] Mathur S, Pilgrim N, Patel SK, Okal J, Mwapasa V, Chipeta E, Musheke M, Mahapatra B, Pulerwitz J. HIV vulnerability among adolescent girls and young women: a multi-country latent class analysis approach. Int J Public Health. 2020 May;65(4):399-411. doi: 10.1007/s00038-020-01350-1. Epub 2020 Apr 9. PMID 32270233
- [Background] Mathur S, Okal J, Musheke M, Pilgrim N, Kishor Patel S, Bhattacharya R, Jani N, Matheka J, Banda L, Mulenga D, Pulerwitz J. High rates of sexual violence by both intimate and non-intimate partners experienced by adolescent girls and young women in Kenya and Zambia: Findings around violence and other negative health outcomes. PLoS One. 2018 Sep 13;13(9):e0203929. doi: 10.1371/journal.pone.0203929. eCollection 2018. PMID 30212561